CLINICAL TRIAL: NCT04144257
Title: Role of Microglial Activation and Norepinephrine Transporter Abnormalities in Pathogenesis of MS-related Fatigue
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency)
Responsible Party: Principal Investigator, TARUN SINGHAL, Assistant Professor of Neurology, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019P002356
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — N-fluoroacetyl-N-(2,5-dimethoxybenzyl)-2-phenoxyaniline

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects diagnosed with Multiple Sclerosis (MS) (Experimental): We plan to enroll 12 subjects with multiple sclerosis (6 with relapsing multiple sclerosis and 6 with secondary progressive multiple sclerosis).
  Interventions: Drug: [F-18]PBR06; Drug: [C-11]Methylreboxetine

INTERVENTIONS:
Drug: [F-18]PBR06 — PET radiopharmaceutical. Subjects will undergo [F-18]PBR06-PET (microglial activation).
  Other Names: [18F]PBR06
Drug: [C-11]Methylreboxetine — PET radiopharmaceutical. Subjects will undergo [C-11]MRB-PET (norepinephrine transporter binding).
  Other Names: [C-11]MRB

SUMMARY:
The overarching aim is to assess the role of microglial activation and norepinephrine transporter binding in pathogenesis of MS-related fatigue, using novel Positron Emission Tomography (PET) radiotracers, [F-18]PBR06 and [C-11]MRB.

Specific Aims:

Specific Aim 1: To determine the relationship of cerebral microglial activation, as assessed by [F-18]PBR06 PET, with MS-related fatigue.

Specific Aim 2: To determine the relationship of norepinephrine transporter (NET) binding, as assessed by [C-11]MRB PET, with MS-related fatigue.

Specific Aim 3: To determine the relationship of microglial activation and NET binding, with grey matter pathology (lesion load and brain atrophy) assessed using 7T MRI, and evaluate their independent contribution in development of MS-related fatigue.

DETAILED DESCRIPTION:
Design: This is a single center, cross-sectional study of patients with multiple sclerosis, who will each, undergo both, [C-11]MRB-PET (norepinephrine transporter binding) and [F-18]PBR06-PET (microglial activation), in addition to 7 Tesla brain MRIs. Patients will also undergo cross-sectional estimations of blood markers.

Genotype Testing:

Blood sample drawn on the initial screening visit will be used to obtain genomic DNA for genotyping for polymorphism within the TSPO gene on chromosome 22q13.2, using a Taqman assay. High affinity and medium affinity binders will be included while the low affinity binders will be excluded from the study.

PET Scanning:

During the PET scan visits, all women subjects of child bearing age will undergo a stat quantitative serum hCG pregnancy test and only women with a negative test will undergo the radiopharmaceutical injection. The radiotracers will be produced using standardized procedures. At the time of imaging, the subjects will be positioned in the gantry of a high-resolution PET/CT camera. Head alignment will be made, relative to the canthomeatal line, using projected laser lines whose positions are known with respect to the slice positions of the scanner. A head support apparatus will be used to minimize head motion.Dynamic data over 120 minutes for PET quantification will be acquired, according to previously described methods for both tracers.

MRI Scanning:

High resolution MRI scanning will be performed using the 7T Siemens MAGNETOM Terra MRI unit at Brigham & Women's Hospital (BWH).

Serum assays:

Serum measurements for inflammatory markers and relevant neurochemicals will be performed according to established procedures.

Clinical Data

The following non-imaging, clinical data will be obtained:

Modified fatigue Impact Scale (MFIS) Fatigue Severity Status Scale (FSSS) Expanded Disability Status Scale (EDSS) Timed 25-feet walk (T25W) MS Functional Composite (MSFC) Symbol digit modalities test (SDMT) MSQOL-54 scale (QOL) Pittsburgh Sleep Quality Index (PSQI) Beck's Depression Inventory (BDI) Center for Epidemiological Studies-Depression Scale (CES-D) Hospital Anxiety and Depression Scale (HADS)

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting the definition for RRMS or SPMS by International Panel (2017 McDonald) Criteria.
* We will recruit patients with RRMS, recently diagnosed in the last 2 years. There will be no disease modifying therapy restrictions for RRMS or SPMS patients.
* Male and female subjects age 18 to 60 years.
* Patients able to withhold medication that may interfere with C-11[MRB] radiotracer uptake for 24 hours before the scan.

Exclusion Criteria:

* Relapse/Corticosteroid treatment in the past 4 weeks to avoid transient effects on imaging
* Individuals with a known alternate neurologic disorder, previous head injury, or substance abuse.
* Individuals with bipolar disease and schizophrenia
* Concurrent medical conditions that contraindicate study procedures.
* Women who are pregnant or nursing. Also, any woman who is seeking to become pregnant or suspects she is pregnant will be excluded from enrollment.
* Claustrophobia
* Non-MRI compatible implanted devices
* Low affinity binders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Standardized Uptake Value (SUV)/Standardized Uptake Value Ratio (SUVR) | Baseline
  PET outcome measure

SECONDARY OUTCOMES:
Modified Fatigue Impact Scale (MFIS) | Baseline
  Clinical outcome measure; Physical subscale range: 0-36; Cognitive subscale range: 0-40; Psychosocial subscale range: 0-8; Total MFIS Score scale range (Subscales Summed): 0-84; Higher values represent worse outcomes.
Binding Potential (BPnd) | Baseline
  PET outcome measure
MRI grey matter lesional load/brain atrophy | Baseline
  MRI outcome measure
Tissue Volume of distribution (Vt)/Distribution Volume Ratios (DVR) | Baseline
  PET outcome measure
MRI global/regional volumetrics | Baseline
  MRI outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Singhal, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Partners MS Center, 60 Fenwood Road, Boston, Massachusetts, United States